CLINICAL TRIAL: NCT00513591
Title: Duke Autoimmunity in Pregnancy Registry
Acronym: DAP Registry
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00000756
Record Dates: First submitted 2007-08-06; First posted 2007-08-08 (Estimated); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: Pregnancy; Systemic Lupus Erythematosus; Cutaneous Lupus; Rheumatoid Arthritis; Sjogren's Syndrome; Scleroderma
Keywords: Pregnancy; Lupus (systemic lupus erythematosus or cutaneous lupus); Rheumatoid Arthritis; Sjogren's Syndrome; Scleroderma
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Arthritis, Rheumatoid; Sjogren's Syndrome; Scleroderma, Diffuse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be collected and stored for future analysis.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: Women with lupus
- 2: Health women who are matched to women with lupus by age and race
- 3: Women with other autoimmune diseases

SUMMARY:
It is difficult to predict how a women with an autoimmune disease will do during pregnancy. Some women will improve, others will worsen. Some pregnancies progress normally and others become very complicated.

The Duke Autoimmunity in Pregnancy (DAP) Registry will enroll women with autoimmune diseases, such as lupus, rheumatoid arthritis, scleroderma, and Sjogren's syndrome who wish to become, or already are, pregnant. We will follow these women throughout pregnancy to better understand how their autoimmune disease affects their pregnancy, and vice versa.

DETAILED DESCRIPTION:
Women with a systemic autoimmune disease that would be followed by a rheumatologist will be included in this study.

All women will be seen every 4-6 weeks throughout pregnancy. At each visit, women will complete a questionnaire, the physician will determine the current level of disease activity, and a blood sample will be taken. For women with lupus and healthy women, and additional visit will occur at the start of the 3rd trimester for a closer evaluation of predictors of preterm birth.

This is not an intervention study. Women will not be given experimental medication. All recommendations for treatment and monitoring will be made based on the best available data with input from the treating obstetrician.

Women in this Registry are not required to be seen by Duke Obstetrics nor to deliver at a Duke Hospital.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Desire for pregnancy within 6 months or currently pregnant
* Women with systemic autoimmune disease, including:

  * Lupus (systemic lupus erythematosus or cutaneous lupus)
  * Antiphospholipid Syndrome or positive antiphospholipid antibodies
  * Rheumatoid Arthritis
  * Scleroderma (systemic sclerosis)
  * Sjogren's Syndrome
  * Inflammatory Arthritis (including Psoriatic Arthritis and Ankylosing Spondylitis)
  * Undifferentiated Connective Tissue Disease (UCTD)
  * Vasculitis
  * Myositis (Polymyositis or Dermatomyositis)
  * Positive Ro/SSA or La/SSB antibodies

Exclusion Criteria:

* Unable to speak English
* Unable to provide informed consent
* Unable to travel to Duke University for follow-up visits

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant women with autoimmune disease.
Sampling Method: Non-Probability Sample
Enrollment: 513 (Actual)
Dates: Start 2007-08; Primary Completion 2018-11-19 (Actual); Study Completion 2018-11-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Megan E. B. Clowse, MD, MPH, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- See also: The Duke Lupus Clinic website — http://www.dukehealth.org/locations/duke_lupus_clinic